CLINICAL TRIAL: NCT07030075
Title: SURVEILLANCE, ASSESSMENT AND DETECTION OF INFLUENZA ASSOCIATED RESPIRATORY INFECTIONS IN HIV POSITIVE AND NEGATIVE INDIVIDUALS IN LUSAKA, ZAMBIA
Status: Recruiting | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: 5955-2024
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Influenza; RSV; COVID - 19
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background and rationale:The World Health Organisation (WHO), estimates influenza global deaths at 290,000 to 650,000 annually. Although influenza is mostly associated with upper respiratory tract infections (URTIs), its role in lower respiratory tract infections (LRTIs) and the associated poor clinical outcomes have been overlooked in sub-Saharan Africa. A study conducted in eight SSA countries estimated that 8.2% of cases and 2.8% of deaths from LRTIs were due to primary infection with influenza. Pneumonia and influenza-associated illness are responsible for 8.5% of respiratory deaths in Zambia. However, in routine practice, testing to distinguish between bacterial and viral etiology of RTIs is seldom done outside sentinel surveillance due to the high cost and lack of available testing options. This consequently underestimates viral RTIs in the population. It is particularly important to diagnose flu early on in vulnerable populations so that they receive timely and appropriate medical care. Although Zambia is a high HIV burden country with a prevalence of 11%, there is presently no study that has described the burden of influenza in the HIV positive population. This research study will address gaps in current scientific knowledge, providing key insights about the prevalence, circulating types, seasonality and associated clinical outcomes of influenza, RSV and SARS-CoV-2 infection in Zambia in the post COVID-19 era.

Objectives Primary To determine the prevalence of influenza (A and/or B) infections in a high HIV burden setting in Lusaka, Zambia over one or more influenza seasons.

Secondary

1. To determine the prevalence of influenza co-infection with RSV and/or SARS-CoV-2
2. To determine the clinical outcomes of influenza (A and/or B) infection among Zambian adults, with and without co-infection with RSV and COVID-19, by HIV and COVID-19 vaccination status.
3. To evaluate the accuracy and yield of aerosol-based sampling for diagnosis of respiratory viruses (influenza, SARS-CoV-2, and RSV) compared to nasal/ nasopharyngeal swabs, for rapid diagnosis of infection among symptomatic individuals in Zambia.
4. To evaluate the acceptability of exhaled breath aerosol (XBA) sampling for diagnosis and screening of respiratory infections of pandemic potential.

Study design and participants:

Primary objective and secondary objective 1:

Cross sectional surveillance study of individuals presenting with flu-like symptoms at two first level hospitals in Lusaka, Zambia. Recruitment of 594 participants will be done over the study period and participants will include both males and females presenting with 2-7 days of flu-like symptoms, able to provide informed consent, aged ≥18 years, with a known HIV status or willing to be tested, with a known COVID 19 vaccination status and available for symptom follow-up.

Secondary objective 2:

Prospective follow up of participants enrolled in aim 1 for 14 days will be done to document clinical symptom progression and outcomes. Appropriate care will be provided to all participants within routine care services.

Secondary objective 3 & 4:

Mixed methods approach. All patients enrolled under aim 1 will be requested to provide in addition to the routine nasopharyngeal sample, an aerosol-based sample for diagnostic accuracy and yield evaluation. We will also conduct an investigator-administered questionnaire to ascertain end-user experience and preferences for either sampling method.

Location Zambia (Kanyama and Chawama sub-districts) Duration April 2025 to November 2026 (Participant enrolment duration)

ELIGIBILITY:
Inclusion Criteria:

* i. age ≥18 years old ii. presenting with flu-like symptoms or acute respiratory infection with ≥2 to 7 days history of cough and /or sore throat and fever, +/- sneezing, +/- congestion, +/- myalgia, +/- fatigue, +/- wheezing, shortness of breath)[55-57] iii. willing to share their HIV status or be tested iv. willing to share their COVID-19 vaccination status v. able and willing to give informed consent vi. willing to provide a nasal/ nasopharyngeal sample for testing as part of standard of care vii. willing to provide exhaled breath aerosol samples i.e. wear a mask and provide a breath sample viii. willing to fill a symptoms diary card for symptom tracking for 7 days ix. agree to be followed-up and attend study visits up to two weeks after study entry

Exclusion Criteria:

* i. individuals who are unwilling to provide any reference standard samples such as the nasopharyngeal swabs ii. those with symptoms for >7 days, or iii. those unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons encountered at the facility entry points will be informed of the study through sensitization activities. Entry points will include the outpatient departments (OPD), emergency room, antiretroviral therapy (ART) clinics, chest clinics, and maternal and child health (MCH) clinics. All adults over the age of 18 years old presenting with flu-like symptoms will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 594 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence | 18months
  Proportion of participants with a positive test (Influenza, RSV or COVID) over the total number of study participants

CONTACTS AND LOCATIONS:
Locations (2):
- Zambia (2):
  - Chawama 1st level Hospital, Lusaka, Lusaka Province
  - Kanyama 1st Level Hospital, Lusaka, Lusaka Province